CLINICAL TRIAL: NCT04494386
Title: Phase 1/2a Study of Umbilical Cord Lining Stem Cells (ULSC) in Patients With ARDS Due to COVID-19
Brief Title: Umbilical Cord Lining Stem Cells (ULSC) in Patients With COVID-19 ARDS
Acronym: ULSC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Restem, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ULSC-CV-01
Record Dates: First submitted 2020-07-24; First posted 2020-07-31 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Covid19; Corona Virus Infection; SARS-CoV Infection; ARDS; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ULSC in Phase 1 Open Label (Experimental): Intravenous (IV) infusion of ULSC in 20 patients with COVID-19 ARDS:
  In Phase 1, two separate cohorts per group will receive either a single dose (one infusion) or repeat dose regimen (two infusions separated by 48-hour interval). The first cohort enrolled will receive the single dose; the next cohort enrolled will be administered the repeat dose regimen.
  Interventions: Biological: Umbilical Cord Lining Stem Cells (ULSC)
- ULSC in Phase 2a Randomized (Experimental): Intravenous (IV) infusion of ULSC in 30 patients with COVID-19 ARDS:
  In Phase 2a, 30 patients assigned ULSC will receive either a single dose (one infusion) or repeat dose regimen (two infusions separated by 48-hour interval). The ULSC dosing regimen will be chosen based on Phase 1 data of safety and tolerability.
  Interventions: Biological: Umbilical Cord Lining Stem Cells (ULSC)
- Placebo in Phase 2a Randomized (Placebo Comparator): Intravenous (IV) infusion of carrier control in 10 patients with COVID-19 ARDS:
  In Phase 2a, 10 patients assigned Placebo will receive either single dose (one infusion) or repeat dose (two infusions separated by 48-hour interval) of carrier control; the dosing regimen will correspond to that of the experimental arm.
  Interventions: Other: Placebo (carrier control)

INTERVENTIONS:
Biological: Umbilical Cord Lining Stem Cells (ULSC) — IV infusion of allogeneic ULSC (100 million cells per dose) in sterile saline for injection
  Other Names: Umbilical Cord Lining Stem Cells (ULSC), type of mesenchymal stem cells (MSC) derived from single donor umbilical cord tissue for allogeneic use
  Arms: ULSC in Phase 1 Open Label; ULSC in Phase 2a Randomized
Other: Placebo (carrier control) — IV infusion of carrier control consisting of sterile saline for injection
  Arms: Placebo in Phase 2a Randomized

SUMMARY:
ULSC-CV-01 is a clinical trial that comprises both Phase 1 and Phase 2a, which will be conducted sequentially. This trial will evaluate the safety and potential efficacy of allogeneic Umbilical Cord Lining Stem Cells (ULSC), which are a type of umbilical cord tissue derived mesenchymal stem cells (MSC), with intravenous (IV) administration in hospitalized patients with acute respiratory distress syndrome (ARDS) due to COVID-19.

DETAILED DESCRIPTION:
The Phase 1, open-label, non-controlled trial in this study will investigate the safety of intravenous (IV) infusion of ULSC in a total of 20 patients with COVID-19-related ARDS that will include patients that are not intubated and not on a ventilator (NV) and patients that are intubated and on a ventilator (V) for respiratory support. Separate cohorts of each group (NV and V) will receive either a single dose (one infusion) or repeat dose (two infusions separated by 48-hour interval).

The Phase 2a randomized and placebo-controlled trial in this study will investigate the potential efficacy of IV infusion of ULSC in a total of 40 patients with COVID-19-related ARDS that will all be EITHER NV or V; the determination of that eligibility criterion and the ULSC dosing regimen will be based on Phase 1 data of safety and tolerability. Phase 2a will evaluate EITHER single dose (one infusion) or repeat dose (two infusions separated by 48-hour interval). The randomization will be 3:1 with 30 patients receiving investigational product (ULSC) and 10 patients receiving placebo (carrier control).

ELIGIBILITY:
Inclusion Criteria:

1. Adult, male or female, age ≥18 years old
2. Diagnosis of the presence of the COVID-19 agent with confirmation of COVID-19 by standard reverse transcriptase polymerase chain reaction (RT-PCR) or equivalent test.
3. Patient with diagnosis of COVID-related ARDS, classified as either:

   * Not requiring mechanical ventilation (NV) or
   * Requiring mechanical ventilation (V).

   According to Berlin Definition of Acute Respiratory Distress Syndrome (ARDS), patients will be categorized based on degrees of hypoxemia [arterial partial pressure of oxygen (PaO2)/oxygen concentration (FiO2)]:
   * Mild ARDS: 200 mm Hg < PaO2/FIO2 ≤ 300 mm Hg
   * Moderate ARDS: 100 mm Hg < PaO2/FIO2 ≤ 200 mm Hg
   * Severe ARDS: PaO2/FIO2 ≤ 100 mm Hg
4. Patient who has exhibited deterioration in condition during the past 72 hours prior to the informed consent.
5. Patient receiving standard of care in-hospital therapy, including appropriate critical oxygenation, fluid, and hemodynamic support as indicated clinically.
6. Patient or responsible family member or surrogate signs informed consent.

Exclusion Criteria

1. Hypersensitivity to study product components. History of hypersensitivity to dimethyl sulfoxide (DMSO).
2. Active cancer or prior diagnosis of cancer within the past year; however, patients with basal and squamous cell cancer of skin will not be excluded.
3. Organ transplant recipient.
4. Chronic renal failure being treated by renal replacement therapy (dialysis) before development of COVID-19.
5. Any other condition that, in the judgment of the Investigator or Sponsor, would be a contraindication to enrollment, study product administration, or follow-up.
6. Pregnancy or lactation; a negative pregnancy test between screening and day 1 (before administration of treatment) will be required of women with childbearing potential, and they will be advised of the requirement to use an effective means of contraception. A woman is considered to be of childbearing potential unless she is postmenopausal and without menses for 12 months or without a uterus and/or both ovaries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLT) | 24 hours
  Number of subjects with a DLT event during or within 24 hours after ULSC infusion
  [Dose Limiting Toxicities are treatment-emergent suspected adverse reactions graded as severe, such as severe infusion-related hypersensitivity toxicities of grade ≥3, and any treatment-emergent serious adverse event (SAE) will be investigated to determine if DLT.]
Incidence of Dose Limiting Toxicity (DLT), suspected adverse reaction (SAR), or serious adverse event (SAE) | 1 week
  Number of subjects with a DLT event, suspected adverse reaction, or any serious adverse event (SAE) within 1 week of each ULSC infusion
Treatment-emergent adverse events (AE) and serious adverse events (SAE) | 1 month
  Treatment-emergent adverse events (AE; incidence, grade, and assessment of relatedness or causality) and serious adverse events (SAE) during the study up to 1-month follow-up
Treatment-emergent adverse events (AE) and serious adverse events (SAE) | 12 months
  Treatment-emergent adverse events (AE; incidence, grade, and assessment of relatedness or causality) and serious adverse events (SAE) during the study and up to the 12-month follow-up

SECONDARY OUTCOMES:
Levels of COVID-19 related ARDS as defined by the Berlin Definition of ARDS | 1 month
  Times to transitions between levels of COVID-19 related ARDS as defined by the Berlin Definition of ARDS
Changes from baseline pulse oximetric saturation SpO2/FiO2 ratio or arterial oxygen pressure pAO2/FiO2 ratio | 1 month
  Changes in SpO2/FiO2 ratio or pAO2/FiO2 ratio compared to baseline, measured daily at a minimum; oxygenation index daily when on ventilator
Number of ventilator-free days (VFD) | 1 month
  Number of ventilator-free days (VFD) in period of 1 month from study treatment
Changes in Complete Blood Count (CBC) with differential from baseline | 1 month, 2 months, 3 months, 6 months, and 12 months
  Changes in CBC with differential from baseline to 1 month, 2 months, 3 months, 6 months, and 12 months after study treatment
Changes in levels of blood glucose (mg/dL) from baseline | 1 month, 2 months, 3 months, 6 months, and 12 months
  Changes in blood glucose (mg/dL) from baseline to 1 month, 2 months, 3 months, 6 months, and 12 months after study treatment
Changes in levels of sodium (mEq/L) from baseline | 1 month, 2 months, 3 months, 6 months, and 12 months
  Changes in levels of sodium (mEq/L) from baseline to 1 month, 2 months, 3 months, 6 months, and 12 months after study treatment
Changes in levels of potassium (mEq/L) from baseline | 1 month, 2 months, 3 months, 6 months, and 12 months
  Changes in levels of potassium (mEq/L) from baseline to 1 month, 2 months, 3 months, 6 months, and 12 months after study treatment
Changes in levels of blood urea nitrogen (BUN; mg/dL) from baseline | 1 month, 2 months, 3 months, 6 months, and 12 months
  Changes in levels of blood urea nitrogen (BUN; mg/dL) from baseline to 1 month, 2 months, 3 months, 6 months, and 12 months after study treatment
Changes in levels of alanine transaminase (ALT; U/L) from baseline | 1 month, 2 months, 3 months, 6 months, and 12 months
  Changes in levels of alanine transaminase (ALT; U/L) from baseline to 1 month, 2 months, 3 months, 6 months, and 12 months after study treatment
Change in Urinalysis (UA) from baseline | 1 month
  Change in Urinalysis (UA) at baseline and 1 month after study treatment to assess for presence and qualitative proteinuria

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Miami Baptist Hospital, Miami, Florida
  - Sanford Research, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No